CLINICAL TRIAL: NCT06857838
Title: Myocardialbridge Bypass Graft Surgery Efficacy Verification
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xi'an International Medical Center Hospital (Other)
Responsible Party: Principal Investigator, Wang zhen, Principal Investigator, Xi'an International Medical Center Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XianInternationalMCH
Record Dates: First submitted 2025-02-20; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Myocardial Bridge of Coronary Artery; Myocardial Bridge; Myocardial Bridging; Myocardial Infarction; Myocardial Ischemia; Pectoris, Stable Angina; Sudden Cardiac Death; Bypass Graft Stenosis; Bypass Graft Occlusion; Bypass Graft Thrombosis
MeSH Terms: conditions — Myocardial Bridging; Myocardial Infarction; Myocardial Ischemia; Angina, Stable; Death, Sudden, Cardiac

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- MyocardialBridge Bypass Graft (Experimental): The patients with deep(depth>2mm) and long-segement(length>25mm) of myocardialbridge receiving myocardialbridge bypass graft surgery(MBBG)，fulfilling the following criteria: 1.presenting with pectoris angina that cannot be effectively relieved by maximum guideline-directed drug therapy; 2. No atherosclerotic plaque or merely mild atherosclerotic stenosis is detected at the proximal or entry of the myocardialbridge confirmed by coronory artery angiography.
  Interventions: Procedure: MBBG
- Myocardialbridge CABG (Active Comparator): The patients with deep(depth>2mm) and long-segement(length>25mm) of myocardialbridge will be allocated to receive myocardialbridge bypass graft surgery(MBBG)，when fulfilling the following criteria: 1.presenting with pectoris angina that cannot be effectively relieved by maximum guideline-directed drug therapy; 2. The moderate-to-severe atherosclertotic stenosis is detected at the proximal or entry of the myocardialbridge confirmed by coronory artery angiography.
  Interventions: Procedure: MB CABG
- Myocardioalbridge Unroof (Active Comparator): The patients with superficial type(depth<2mm) and short-segement(length<25mm) of myocardial bridge will be allocated to receive "unroof" surgery，when fulfilling the following criteria: 1.presenting with pectoris angina that cannot be effectively relieved by maximum guideline-directed drug therapy; 2. No atherosclerotic plaque or merely mild atherosclerotic stenosis is detected at the proximal or entry end of the myocardialbridge confirmed by coronory artery angiography.
  Interventions: Procedure: MB unroof

INTERVENTIONS:
Procedure: MBBG — The patients with deep(depth>2mm) and long-segement(length>25mm) of myocardialbridge receiving myocardialbridge bypass graft surgery(MBBG)，fulfilling the following criteria: 1.presenting with pectoris angina that cannot be effectively relieved by maximum guideline-directed drug therapy; 2. No atherosclerotic plaque or merely mild atherosclerotic stenosis is detected at the proximal or entry of the myocardialbridge confirmed by coronory artery angiography.
  Arms: MyocardialBridge Bypass Graft
Procedure: MB CABG — The patients with deep(depth>2mm) and long-segement(length>25mm) of myocardialbridge receiving myocardialbridge bypass graft surgery(MBBG)，fulfilling the following criteria: 1.presenting with pectoris angina that cannot be effectively relieved by maximum guideline-directed drug therapy; 2. The moderate-to-severe atherosclerotic stenosis is detected at the proximal or entry of the myocardialbridge confirmed by coronory artery angiography.
  Arms: Myocardialbridge CABG
Procedure: MB unroof — The patients with superficial type(depth<2mm) and short-segement(length<25mm) of myocardial bridge will be allocated to receive myocardialbridge "unroof" surgery，when fulfilling the following criteria: 1.presenting with pectoris angina that cannot be effectively relieved by maximum guideline-directed drug therapy; 2. The MB was superficial and short confirmed by coronory artery CT angiography.
  Arms: Myocardioalbridge Unroof

SUMMARY:
Myocardial Bridge Bypass Graft surgery is introduced to relieve the unmedical symptoms of patients with long-segment or deep myocardial bridge, clinical outcomes will be collected to verify the effectiveness of the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with myocardialbridge requiring drug therapy or surgical intervention.

Exclusion Criteria:

* patients with myocardialbridge not requiring drug therapy or surgical intervention, or unwilling to be enrolled for any reason

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
All-Cause Mortality | Up to 240 months
Rate of counduit patency | Up to 180 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Wang, Doctorate, Principal Investigator — Xi'an International Medical Center Hospital Affiliated To Northwest University; Jinzhou Zhang, Doctorate, Study Director — Xi'an International Medical Center Hospital Affiliated To Northwest University; Jinzhou Zhang, Doctorate, Study Chair — Xi'an International Medical Center Hospital Affiliated To Northwest University
Locations (1):
- Xi'an International Medical Center Hospital Affiliated TO Northwest University, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Zhang JZ, Zhu GY, Zhang Y, Bai LJ, Wang Z. Myocardial Bridge Bypass Graft: A Novel Surgical Procedure for Extensive Myocardial Bridges. Ann Thorac Surg. 2021 Aug;112(2):e115-e117. doi: 10.1016/j.athoracsur.2020.11.055. Epub 2021 Jan 20. PMID 33482166
- See also: The report of the preliminary short term clinical results of MBBG surgery for the first time in the world — http://pubmed.ncbi.nlm.nih.gov/33482166/